CLINICAL TRIAL: NCT05200819
Title: Incidence and Predictors of Acute and Chronic Complications in Patients With Diabetes and Severe COVID-19
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Professor of Internal Medicine Metabolism, Endocrinology and Diabetes Vice Chair of Clinical Research Department of Internal Medicine Associate Director, Clinical Research, Mentoring and Development, Elizabeth Weiser Caswell Diabetes Institute, University of Michigan
Other Study IDs: HUM00186076
Record Dates: First submitted 2022-01-17; First posted 2022-01-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Covid19; Diabetes Mellitus
Keywords: Covid19; Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19 Patients: Patients who have survived COVID-19 infection, including those included in the Michigan Medicine COVID-19 Cohort (M2C2) will be eligible to participate.

SUMMARY:
All surviving patients of the Michigan Medicine COVID-19 Cohort (M2C2, PI: Hayek) that were admitted to the University of Michigan for severe COVID-19 disease are eligible for this study. Investigators had prior approval from the Institutional Review Board (IRB) to collect the baseline blood and urine samples of these participants. Initial analysis on those samples are ongoing. In preliminary analysis of these patients a significantly higher risk for severe acute complications in patients with diabetes compared to those without diabetes was observed. The study will also enroll people following documented COVID-19 infection, regardless of whether or not they were hospitalized. The goal of the study is to understand what drives the increased risk of severe acute COVID-19 complications as well as to understand the long term sequelae of COVID-19 infection in patients with diabetes. The objectives of this study are to invite surviving M2C2 participants as well as others who have survived COVID-19 infection for an in-person visit, to measure biomarkers of inflammation and kidney, nerves, heart and blood vessels damage. participants will also be comprehensively phenotyped for diabetic complications outcomes, diabetes kidney disease, diabetes neuropathy and cardiovascular disease. Participants will be asked to fill out questionnaires to assess psychosocial metrics. The rationale is that correlating markers of acute hyperinflammation (cytokine storm syndrome) at admission in diabetes patients can inform vigilance and care for long term complications in survivors. Completing these studies will generate evidence-based guidelines for mitigating sequelae in diabetes COVID-19 survivors and identify critical psychosocial factors to mitigate psychological harm.

DETAILED DESCRIPTION:
Diabetic patients, particularly those with type 2 diabetes (T2D), are highly susceptible to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) induced adverse outcomes and complications. The massive global T2D burden and high COVID-19 infection rate is creating large and significantly vulnerable COVID-19 T2D patient populations.

The prevalence of diabetes among admitted COVID-19 infections has varied 20-50% by region.T2D patients are more prone to a severe COVID-19 disease course, marked by dangerous infection-induced adverse outcomes and complications including intensive care unit (ICU) admission, mechanical ventilation use, or death. The clinical experience with patients admitted to the Michigan Medicine COVID-19 Cohort (M2C2, PI: Hayek): 42% of COVID-19 cases had diabetes, and a disproportionally larger fraction, 56%, required ICU admittance and suffered over twice the mortality (22%) compared to non-diabetic (10%) patients. Thus, T2D consistently predisposes COVID-19 patients to poorer prospects, including acute kidney injury, cardiovascular complications and death.

Most T2D patients frequently suffer from comorbidities, including metabolic syndrome (obesity, hypertension), chronic inflammation, and vascular diabetic complications, i.e., diabetic kidney disease (DKD), diabetic neuropathy (DN), and cardiovascular disease (CVD). In the multi-center French Coronavirus SARS-CoV-2 and Diabetes Outcomes (CORONADO) study (n=1,317 diabetic participants, 88.5% T2D), obesity, measured by body mass index (BMI) positively predicted the study primary outcome, tracheal intubation for mechanical ventilation and/or death within 7 days of admission. The presence of micro- and macrovascular complications at admission independently associated with 7-day mortality, as did inflammation [C-reactive protein (CRP)]and liver injury at admission. Thus, T2D patients, through their comorbid conditions, are at an especially dangerous risk of serious COVID-19 infection and death.

The underlying reasons for the T2D patient susceptibility to COVID-19 remains unclear, although there are several theories. One is that COVID-19-induced cytokine storm syndrome (CSS) may superimpose on the chronic inflammation already present in T2D, promoting a vicious cycle of cytokine release and hyperglycemic surges. T2D is characterized by a chronic, low-grade inflammation, which is also a feature of its complications, DKD, DN, and CVD. Importantly, there are no studies stratifying patients by diabetes status to determine whether a biomarker would be especially useful for predicting the clinical course in COVID-19 T2D patients.

It is also becoming clear that COVID-19 survivors may face a lifetime of sequelae. As with acute infection, T2D patients may also be particularly at risk here. Although the pandemic has not yet lasted long enough to measure long term outcomes, the evidence to date suggests a significant burden of new complications. For instance, COVID-19 may aggravate preexisting pathology, including in T2D patients, and multi-organ injury that aggravates tissues already weakened by preexisting diabetic complications. Finally, the COVID-19 pandemic has seen racial health disparities soar. SARS outbreak survivors report long term effects, even years later, including psychological and financial hardship. In addition, given the disparity during the COVID-19 pandemic, racial minorities faced even more hardships. Identifying these psychosocial factors could mitigate long term psychological trauma. The challenges of the long-term consequences of COVID-19 are emerging as a growing number of patients are long-term survivor sequelae. Identifying these COVID-19 patients who experienced serious clinical complications during their inpatient hospitalization and then sequelae after the acute phase, will deliver better long term outpatient care and allow to preemptively screen for new onset and progression in all complications.

ELIGIBILITY:
Inclusion Criteria • Have been diagnosed with COVID-19 and/or admitted with severe COVID19

Exclusion Criteria

• Women who are currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living patients who were hospitalized for COVID-19 infection (Michigan Medicine COVID-19 or M2C2 Cohort) will be invited to participate in this study. In addition, any patient who has survived COVID-19 infection (regardless of whether they were hospitalized) may be enrolled.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Risk-marker signatures for severe COVID-19 disease, longer-term complications in patients surviving COVID-19. | Single visit lasting 2 to 6 hours. Visit will occur within 3 years of COVID-19 diagnosis
  Comprehensively phenotype COVID-19 survivors for vascular outcomes including kidney disease, peripheral and autonomic neuropathy, cardiovascular disease, as well as cognitive disorders and and patient-reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, M.D., Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No